CLINICAL TRIAL: NCT06799104
Title: EFFECT OF PYRAMIDAL TRAINING ON EPICARDIAL FAT FOR CORONARY ARTERY DISEASE PREVENTION
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rawda Mohamed Ahmed Mohamed El Komy, Principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P.T.REC/012/005563
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Coronary Artery Disease; Class I Obesity
Keywords: Pyramidal Training, Epicardial Fat,Coronary artery disease.
MeSH Terms: conditions — Coronary Artery Disease | interventions — Diet, Mediterranean

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group: (Experimental): This group will include 25 patients who will receive pyramidal aerobic training by treadmill for 40 minutes per session (three sessions per week) for (12 weeks) in addition to Mediterranean diet.
  Interventions: Other: Pyramidal training; Other: Mediterranean diet
- Control group (Active Comparator): This group will include 25 patients who will receive Mediterranean diet for (12 weeks).
  Interventions: Other: Mediterranean diet

INTERVENTIONS:
Other: Pyramidal training — Pyramidal training prescription:Mode of exercise: aerobic interval training. Intensity: ranging from 20-80% from THR. Duration: 40 minutes per session.Frequency: Three sessions per week for 12 weeks.
  The course of the program will be 2 sets of pyramidal training with 10 minutes for rest between them. Each set will be 5 levels of incremental and 5 levels of decremental aerobic exercise and each level 2 minutes on a treadmill.
  1. Level one: will be set as a 20% walking of Karvonen formula.
  2. Level two: will be set as a 30% running of Karvonen formula.
  3. Level three: will be set as a 50%running of Karvonen formula.
  4. Level four: will be set as a 70% running of Karvonen formula.
  5. Level five: will be set as a 80% running of Karvonen formula.
  Arms: Experimental group:
Other: Mediterranean diet — Mediterranean diet:
  Meal Composition Main meals consumed daily should be a combination of three elements: cereals, vegetables and fruits, and a small quantity of legumes, beans or other (though not in every meal). Cereals in the form of bread, pasta, rice, couscous or bulgur (cracked wheat) should be consumed as one-two servings per meal. Vegetable consumption should amount to two or more servings per day, in raw form for at least one of the two main meals (lunch and dinner). Fruit should be considered as the primary form of dessert, with one-two servings per meal.

SUMMARY:
To show the effect of pyramidal training for coronary artery disease prevention on:

-Epicardial fat, BMI, Waist circumference (WC), Lipid profile, Quality of life and Mediterranean Diet Adherence.

DETAILED DESCRIPTION:
Back Ground: Coronary heart disease (CHD) is a type of ischemic heart disease characterized by atherosclerotic plaque accumulation in the coronary arteries.Obesity leads to coronary artery disease (CAD) in part through an inflammatory process that accelerates atherosclerotic plaque formation which may start as early as childhood. Epicardial adipose tissue (EAT) is the Visceral adipose tissue (VAT) of the heart .EAT has unique embryologic, anatomic, and histologic features, including smaller adipocytes and higher prevalence of immune cells when compared to subcutaneous adipose tissue (SAT).

Purpose: To show the effect of pyramidal training for coronary artery disease prevention on:

-Epicardial fat, BMI, Waist circumference (WC), Lipid profile, Quality of life and Mediterranean Diet Adherence.

Methods: This study is Randomize Control Trail that will be carried out on 50 females' patients and will be selected from the Outpatient clinics at Pharos University. Patient will be randomly assigned to two groups.

Experimental group:

This group will include 25 patients who will receive pyramidal aerobic training by treadmill for 40 minutes per session (three sessions per week) for (12 weeks) in addition to Mediterranean diet.

Control group:

This group will include 25 patients who will receive Mediterranean diet for (12 weeks).

Results: Data analysis with Independent t-test will be used to compare the baseline parameters between the intervention and control groups. Repeated measures ANOVA will be used to compare the changes in EATT, anthropometrics and lipid levels at the baseline and after 12 weeks between the two groups.

Keywords: Pyramidal Training, Epicardial Fat, Coronary artery disease.

ELIGIBILITY:
Inclusion Criteria:

* Fifty females' patients with class I obesity (BMI 30 to 34.9 kg/m2, Waist circumference > 88 cm).

  * Their age ranges from 30-40 years old.
  * Dyslipidemia and lipid profile as follow (total cholesterol high: 240 mg/dl, HDL less than 40 mg/dl, LDL high: 160-189 mg/dL and triglycerides high: 200-499 mg/dl).
  * All patients will be clinically and medically stable when attending the study.

Exclusion Criteria:

* Patients with conditions will be excluded such as:

  * Musculoskeletal problems.
  * Chronic pulmonary disease.
  * Missed more than two weeks of the program or want to terminate the program.
  * Unstable angina.
  * Acute illness.
  * Uncontrolled cardiac arrhythmia.
  * Decompensated heart failure.
  * Cognitive impairment or mental disorders.
  * Systolic blood pressure higher than 180, and/or diastolic blood pressure over 100mmHg.
  * DVT.
  * Multiple food allergies/intolerances or gastrointestinal difficulties of the prescribed diet.
  * Cancer (have special nutritional and training needs).

Ages: 30 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Epicardial adipose tissue thickness. | 12 weeks
  The echo measurements for EATT will be taken in standard parasternal view in the left lateral decubitus position by an experienced cardiologist, and the mean values between long- and short-axis views will record. The EAT is identify as the echo-free space between the outer wall of the myocardium and the visceral layer of the pericardium. The thickness is measure perpendicularly on the free wall of the right ventricle at end systole in three to ten cardiac cycles

SECONDARY OUTCOMES:
(lipid profile) Blood test | 12 weeks
  Blood sampling will conduct 48 hours before the first training session and 48 hours after the last training session. Participants will instruct to stop eating for at least eight hours prior to the blood sample.
Anthropometric measurements | 12 weeks
  BMI was calculated by dividing body weight (kg) by the square of length (m2). Between 18.5-24.9 kg/m2 , BMI is defined as normal, between 25.0-29.9 kg/m2 as overweight, ≥30 kg/m2 as obesity, and ≥35 as severe obesity. WC was measured from the midpoint of the lateral iliac prominences and the lowest rib while standing. It was high considered as 88 cm and above in women, 102 cm and above in men. Hip circumference was measured around the widest part of the hip, and WHR was calculated by dividing WC (cm) by hip circumference (cm). It was high considered as 0.85 and above in women, 0.90 and above in men
Impact of Weight on Quality of Life-Lite Clinical Trials Version (IWQOL-Lite-CT) | 12 weeks
  The IWQOL-Lite-CT is a 20-item patient-reported outcome (PRO) measure designed to assess the impact of changes in weight on patients' physical and psychosocial functioning. Each item employs a 5-point graded response scale (never, rarely, sometimes, usually, always; or not at all true, a little true, moderately true, mostly true, completely true). In addition to yielding a Total score, the final 20-item IWQOL-Lite-CT includes two primary domains: Physical (7 items) and Psychosocial (13 items)
14-Item Mediterranean Diet Adherence Screener (MEDAS) | 12 weeks
  The MEDAS is a 14-item questionnaire requesting participants to report the habitual frequency of consumption or amount consumed of 12 main components of the MedDiet and two food habits related to the MedDiet. Each of the 14 items is scored 1 or 0, depending on whether participants adhere to each MedDiet component or not. If these conditions were not met, an item was assigned a score of 0. The resulting MEDAS-derived MedDiet score ranged from 0 to 14

CONTACTS AND LOCATIONS:
Overall Officials: Zeinab M Helmy, Professor, Study Chair — Cairo University; Ebtesam N Abdel-Mohsen, PhD, Study Director — Cairo University; Hoda A Saad ELDin, PhD, Study Director — Alexandria University
Locations (1):
- Cairo University, Cairo, Giza Governorate, Egypt